CLINICAL TRIAL: NCT05457829
Title: Doxorubicin Hydrochloride Liposome Combined With Irinotecan (AI Regimen) Versus VIT Regimen in the Treatment of First Relapsed and Refractory Pediatric Rhabdomyosarcoma: a Prospective, Open-label, Randomized Controlled, Multicenter, Phase II Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director of department of pediatric cancer,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PST-01
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Rhabdomyosarcoma, Child
Keywords: Rhabdomyosarcoma; Doxorubicin Hydrochloride Liposome Injection; Irinotecan
MeSH Terms: conditions — Rhabdomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI Regimen (Experimental): Doxorubicin hydrochloride liposome injection combined with Irinotecan
  Interventions: Drug: Doxorubicin Hydrochloride Liposome+Irinotecan
- VIT Regimen (Active Comparator): Temozolomide combined with Irinotecan and Vincristine
  Interventions: Drug: Temozolomide+Irinotecan+Vincristine

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride Liposome+Irinotecan — Q3W, 2 cycles.
  Arms: AI Regimen
Drug: Temozolomide+Irinotecan+Vincristine — Q3W, 2 cycles.
  Arms: VIT Regimen

SUMMARY:
This multicenter, randomized, controlled, open-label, prospective clinical trial was designed to evaluate the efficacy and safety of doxorubicin hydrochloride liposome injection in combination with irinotican (AI regimen) versus VIT regimen in the treatment of first relapsed and refractory pediatric rhabdomyosarcoma.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the objective response rate (ORR) of first relapsed and refractory rhabdomyosarcoma in children after 2 cycles of chemotherapy with AI or VIT regimens. Secondary objectives were to evaluate the disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and safety of AI and VIT regimen in the treatment of relapsed and refractory pediatric rhabdomyosarcoma.

ELIGIBILITY:
Inclusion Criteria

1. 6 months ≤age≤18 years, no gender limitation;
2. The Karnofsky (≥16 years old) or Lansky (< 16 years old) physical status score is at least 50;
3. The expected survival time is not less than 12 weeks;
4. Heart function: A) Cardiac COLOR ultrasound detection LVEF≥ 50%; B) EKG suggests no myocardial ischemia;C) No history of arrhythmia requiring drug intervention before enrollment;
5. Patients who meet the clinical diagnostic criteria and are diagnosed with pediatric rhabdomyosarcoma;
6. Patients who have progressed, relapsed or refractory after first-line treatment (failed to achieve complete or partial response after recent treatment);
7. Measurable lesions (according to RECIST 1.1 standards, CT scan length of tumor lesions ≥10mm, CT scan short diameter of lymph node lesions ≥15mm, measurable lesions have not received radiotherapy, freezing and other local treatments);
8. The patient must fully recover from the acute toxic effects of all previous anticancer chemotherapy: A) Myelosuppressive chemotherapy: at least 21 days after the last myelosuppressive chemotherapy (42 days if nitrosourea was used previously);B) Experimental drug or anticancer therapy other than chemotherapy: not available within the first 28 days of planned initiation of AI or VIT. Complete recovery from clinically significant toxicity of the therapy must be determined;C) Hematopoietic growth factor: at least 14 days after the last administration of long-acting growth factor or 3 days after the last administration of short-acting growth factor;D) Immunotherapy: at least 42 days after completion of any type of immunotherapy (except steroids), such as immune checkpoint inhibitors and tumor vaccines; E) X-ray therapy (XRT) : at least 14 days after local palliative XRT (small mouth); For other substantial bone marrow (BM) irradiation, it must be completed for at least 42 days; F) Stem cell infusion without total body irradiation (TBI) : there is no evidence of active graft-versus-host disease and the transplant or stem cell infusion must be completed at least 56 days after the infusion;
9. Laboratory tests during screening should meet the following conditions: A) Absolute value of neutrophils (ANC) ≥1.5×109/L (if bone marrow invasion, ANC≥1.0×109/L); B) Platelet count (PLT) ≥75×109/L (PLT≥50×109/L for bone marrow invasion); C) Bilirubin (sum of combined + uncombined) ≤ 2.5× upper limit of normal value (ULN) (corresponding to age), patients with confirmed Gilbert's syndrome can be included in the group according to the investigator's judgment; D) Estimated glomerular filtration rate ≥30 mL/min/1.73 m2 or serum creatinine (Cr) ≤ 1.5ULN (calculated according to the standard Cockcroft-Gault formula); E) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN (5 times ULN if liver metastasis is present)
10. Able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits during the study period;
11. The parent/guardian of the child or adolescent subject is capable of understanding, agreeing to, and signing the study Informed consent (ICF) and the applicable child consent form prior to initiating any program-related procedures; Subject is capable of expressing consent with parental/guardian consent (if applicable).

Exclusion criteria

1. Patients who had previously received irinotecan combined with temozolomide and vincristine, or who had progressed after treatment with irinotecan or temozolomide, or who had previously received doxorubicin hydrochloride liposome injection chemotherapy;
2. P450 enzyme-induced anticonvulsants (anticonvulsants affect irinotecan clearance);
3. Previous or concurrent clinical significance of active cardiovascular diseases, including congenital heart disease or pericardial disease, history of heart failure, myocardial infarction, coronary heart disease, heart valvular disease, cardiomyopathy, arrhythmias (including persistent atrial fibrillation, complete left bundle branch block, frequent ventricular premature onset); Or prolonged QT interval (QTc) after current corrected heart rate > 480 ms; Patients with grade III ~ IV cardiac insufficiency according to the New York Heart Association (NYHA) cardiac function classification (age > 3 years) or infant cardiac function standard (age ≤3 years), or left ventricular ejection fraction (LVEF) < 50% as indicated by color doppler echocardiography;
4. Severe chronic skin diseases in the past;
5. Previous allergic asthma or severe allergic disease;
6. Poorly controlled hypertension and diabetes;
7. Have a history of other tumors, except cured cervical cancer or basal cell carcinoma of the skin;
8. Hepatitis B surface antigen positive patients;
9. HIV or syphilis infected patients;
10. Patients who have previously received organ transplants;
11. Uncontrolled and active systemic bacterial, viral or fungal infection;
12. Contraindications to the use of large doses of hormones, such as uncontrolled hyperglycemia, gastric ulcers or mental diseases;
13. Patients who had used doxorubicin at a cumulative dose of ≥450 mg/m2, or epirubicin at a cumulative dose of ≥ 550 mg/m2, or who had used anthracyclines in the past to induce heart disease;
14. Have a history of severe neurological or psychiatric disorders, including epilepsy or autism.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 cycles of chemotherapy（each cycle is 21 days）
  Objective response rate (ORR) after 2 cycles of chemotherapy with AI or VIT regimen, including complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 2 cycles of chemotherapy
  Refers to the percentage of patients with confirmed complete response, partial response, and disease stability in patients with evaluable efficacy.
Progression-free survival (PFS) | From date of radomization unit the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 moths
  Means from the date of enrollment to the date of first disease progression or death from any cause, whichever comes first. If the subject has no disease progression during the trial period, PFS is defined as the last date until the subject's last confirmed progression-free survival.
Overall survival (OS) | From date of radomization unit the date of first documented date of death from any cause, assessed up to 36 moths
  Overall survival (OS) was defined from the date of enrollment to the date of death from any cause.
Adverse events (AE) | Time from the date of enrollment to 30 days after the last dose.
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No